CLINICAL TRIAL: NCT00511290
Title: Measurement of Soluble Factors and Particulate Matter in Induced Sputum and EBC in Inflammatory Diseases of the Lung
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-07-LF-07316-CTIL
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Interstitial Lung Diseases; Occupational Lung Diseases
Keywords: Primary disease or condition being studied: Asthma -COPD-Interstitial Lung Diseases-Occupational Lung Diseases
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no generic names

SUMMARY:
In the present study inflammatory mediators will be isolated in induced sputum and exhaled breath condensate and will be correlated with particulate matter measured in these samples.Particulate matter will be assessed by partcle size distribution method and shape analysis.

The aim of the study is to perform biological monitoring in environmental and occupational diseases in a non invassive fashion.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-80

Exclusion Criteria:

* FEV1 < 75% predicted pO2 < 75

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Fireman Lizy, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel